CLINICAL TRIAL: NCT01739998
Title: Randomized, Double-blind, Controlled Study to Evaluate the Efficacy of Omega 3 Fatty Acids on Different Inflammatory Markers in Obese Subjects With Dietary Intervention for Weight Lost
Brief Title: Health Benefits of Functional Oil (Mega 3 Fatty Acids From Fish Oil) on Obese People
Acronym: NOBO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: NOBO
Record Dates: First submitted 2012-11-27; First posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Functional Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- functional oil (Experimental): Treatment consisted of consuming 5 ml of functional oil [olive oil (4 ml) with omega 3 fatty acids from fish oil (1 ml: 90% omega 3: 75-80% DHA and 10-15% EPA) Orange flavour] during the day by 8 weeks.
  Interventions: Dietary Supplement: functional oil
- Placebo (Placebo Comparator): Treatment consisted of consuming 5 ml of olive oil during the day by 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: functional oil
  Arms: functional oil
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Examine the effects and safety of functional oil (olive oil with omega 3 fatty acids from fish oil) on different inflammatory markers in obese subjects with dietary intervention for weight lost.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from 30 to 75 years old.
* Body mass index (BMI) ≥ 30 kg/m2
* Signed informed consent.

Exclusion Criteria:

* Individuals with special diet due to disease as celiac disease, chronic renal failure, etc.
* Individuals with Diabetes Mellitus insulin dependent.
* Individuals with disorders associated with eating behaviour.
* Individuals with mental disease or low cognitive function.
* Individuals with consumption of drugs to weight lost.
* Individuals treated with drugs whose direct effect is on lipid profile (statins, fibrates, diuretics, corticosteroids or oral anti-inflammatory).
* Individuals with diseases that could be involucrate in weight lost (not controlled hypothyroidism, serious psychiatric illness, etc.)
* Pregnant women or lactating.
* Individuals with recurrent infections.
* Individuals with regular consumption of anti-inflammatory or glucocorticoids.
* Individuals with consumption of oil fish supplements (except if they gave up its consumption 1 month before).
* Individuals with fish allergy.
* Individuals with consumption of more than two fatty fish servers twice a week.
* Individuals with physical problems complying with the recommendations of physical activity and diet indicated.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Inflammatory markers | 2 months
  Inflammatory markers (Adiponectin, fibrinogen, TNFα, PAI-1 and PCR

SECONDARY OUTCOMES:
Anthropometric parameters | 0.1 and 2 months
  Parameters measured were: Weight, Height and waist circumference, muscle mass percentage (MM%), fat mass percentage (FM%).
Lipid profile | 0.1 and 2 months
  Parameters measured were: Cholesterol, LDL-Cholesterol, HDL-Cholesterol, Triglycerides, ApoB, ApoA1 and plasma free fatty acids.
Hormonal Parameters | 0.2 months
  Parameters measured were: Leptin and ghrelin
Oxidative Stress Parameters | 0 and 2 months
  Parameters measured were: plasma antioxidant capacity (FRAP, ferric reducing antioxidant power) and lipidic peroxidation (TBARS, thiobarbituric acid reactive substances assay).
Glucosa Metabolism | 0, 1 and 2 months
  Parameters measured were: glucose, basal insulin, HbA1c (in diabetic patients), HOMA index (glucemic insulin sensitivity index was calculated using the formula: HOMA-IR = fasting glucose (mmol/l)/fasting immunoreactive insulin (mU/ml)/22•5).
Depression Test | 0 and 2 months
  Parameters measured were: Beck Depression Inventory (BDI).
Motivation and Satiety Parameters | 0 and 2 month
  Parameters measured were: Visual analogue scale to assess motivation and satiety to eat.
Adeherence and Tolerance parameters | up to 2 months
  Questionnaire of adherence and tolerance to the product.